CLINICAL TRIAL: NCT06920017
Title: Demographic Data and Clinical Presentation of Pediatric Uveitis Patients in Upper Egypt.
Brief Title: Demographic Data and Clinical Presentation of Pediatric Uveitis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hasnaa Salah Ebrahim Abo Elyuon, Dr, Assiut University
Other Study IDs: Pediatric Uveitis
Record Dates: First submitted 2025-03-13; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Pediatric Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To describe and analyze the demographics, Clinical characteristics, etiology, and visual outcomes of pediatric uveitis cases attending the outpatient clinic of Ophthalmology department, Assiut University Hospital.

DETAILED DESCRIPTION:
Uveitis is a form of eye inflammation that affects the middle layer of tissue in the eye wall (uvea).

It is the third leading cause of blindness worldwide .Uveitis is more common in adults; however, children comprise 2.2% to 21.6% of patients in various studies.Despite a lower incidence of uveitis in children, the rate of visual loss may be worse than that of adults . The onset of uveitis in children is often insidious and is only discovered during routine screening.The lack of significant symptoms and delayed presentation to an ophthalmologist leads to morbidity and a decrease in visual acuity . The length of time between the diagnosis of uveitis and the referral to a tertiary eye center is strongly correlated with the complications rate and degree of visual impairment.

Uveitis is classified according to the International Uveitis Study Group criteria based on the anatomical location of the inflammation and is categorized as anterior, intermediate, Posterior or panuveitis. It is also described based on clinical onset, duration and course.

Some uveitis syndromes are unique to children, such as juvenile idiopathic arthritis (JIA), Kawasaki syndrome, Familial Juvenile Systemic Granulomatosis and Tubulointerstitial Nephritis-Uveitis syndrome. Other conditions are more prevalent in the pediatric population due to environmental factors such as trematode induced uveitis.

Due to the lack of epidemiological studies on the demographic and Clinical Characteristics of pediatric uveitis in Upper Egypt. This study aims to improve diagnosis, management, and treatment strategies tailored to the population.

ELIGIBILITY:
Inclusion Criteria:

* Uveitis patients <18 years old
* must be able to participate in the study.

Exclusion Criteria:

* Age over 18 years.
* Patients with post pentrating ocular trauma.
* Patients whose legal guardians are unwilling to participate in the study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Distribution of uveitis subtypes. | Baseline
Differences by age, gender, or ethnicity. | Baseline
Prevalence of systemic associations. | Baseline
Prevalence of Visual outcomes. | Baseline
Prevalence of complications rate. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Sharaf El Din Abd El Rahim, professor, Study Director — Assiut University; Mohmed Gamal Ahmed Saleh, Assistant Professor, Study Director — Assiut University; Eslam Mohamed Mohamed Goda, Lecturer, Study Director — Assiut University

REFERENCES:
- [Background] .Nussenblatt RB, Whitcup SM. Uveitis: Fundamentals and Clinical Practice, 4th edition. Mosby, 2010
- [Background] Jabs DA, Nussenblatt RB, Rosenbaum JT; Standardization of Uveitis Nomenclature (SUN) Working Group. Standardization of uveitis nomenclature for reporting clinical data. Results of the First International Workshop. Am J Ophthalmol. 2005 Sep;140(3):509-16. doi: 10.1016/j.ajo.2005.03.057. PMID 16196117
- [Background] American Academy of Ophthalmology meeting (Uveitis and Ocular Inflammation section), October 25, 2004; New Orleans, Louisiana
- [Background] Rahimi M, Oustad M, Ashrafi A. Demographic and Clinical Features of Pediatric Uveitis at a Tertiary Referral Center in Iran. Middle East Afr J Ophthalmol. 2016 Jul-Sep;23(3):237-40. doi: 10.4103/0974-9233.186096. PMID 27555706
- [Background] Chan NS, Choi J, Cheung CMG. Pediatric Uveitis. Asia Pac J Ophthalmol (Phila). 2018 May-Jun;7(3):192-199. doi: 10.22608/APO.2018116. Epub 2018 Apr 23. PMID 29682916
- [Background] Cunningham ET Jr. Uveitis in children. Ocul Immunol Inflamm. 2000 Dec;8(4):251-61. doi: 10.1076/ocii.8.4.251.6459. PMID 11262655
- [Background] Rosenberg KD, Feuer WJ, Davis JL. Ocular complications of pediatric uveitis. Ophthalmology. 2004 Dec;111(12):2299-306. doi: 10.1016/j.ophtha.2004.06.014. PMID 15582090
- [Background] Edelsten C, Reddy MA, Stanford MR, Graham EM. Visual loss associated with pediatric uveitis in english primary and referral centers. Am J Ophthalmol. 2003 May;135(5):676-80. doi: 10.1016/s0002-9394(02)02148-7. PMID 12719076
- [Background] Azar D, Martin F. Paediatric uveitis: a Sydney clinic experience. Clin Exp Ophthalmol. 2004 Oct;32(5):468-71. doi: 10.1111/j.1442-9071.2004.00864.x. PMID 15498056
- [Background] Kump LI, Cervantes-Castaneda RA, Androudi SN, Foster CS. Analysis of pediatric uveitis cases at a tertiary referral center. Ophthalmology. 2005 Jul;112(7):1287-92. doi: 10.1016/j.ophtha.2005.01.044. PMID 15921752
- [Background] Benezra D, Cohen E, Maftzir G. Patterns of intraocular inflammation in children. Bull Soc Belge Ophtalmol. 2001;(279):35-8. PMID 11344713